CLINICAL TRIAL: NCT00249886
Title: Discontinuation Study Of Citalopram (Antidepressant) in Depressed Adolescents
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISRCTN42386710
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2005-11

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Citalopram

INTERVENTIONS:
Drug: Citalopram

SUMMARY:
The purpose of the study is to evaluate whether it is advantageous for adolescents who have recovered from depression after a 6 to 12 week course of antidepressant treatment to stay on the treatment a further 6 months or is it just as helpful to stop the medication after recovery.

The hypothesis is that adolescents with major depression who recover from the 6 to 12 week trial of citalopram will be less likely to have a recurrence of depression over a 6 month period if continued on the citalopram as compared to those who discontinue the medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major Depression.
* Age 13-18.
* A score of > 16 on the 17 item Hamilton Depression Scale or a score of > 12 on the 17 items plus a score of >7 on the atypical items.
* Males and females.
* Outpatient at initiation of double blind treatment phase.
* Ability to give informed consent.

Exclusion Criteria:

* Past or current hypomanic or manic episode.
* Currently meets criteria for a Conduct Disorder.
* Current psychotic symptoms.
* Substance dependence in the last 3 months.
* Significant medical condition that would contraindicate the use of an antidepressant.
* Pregnancy
* Past treatment with Citalopram for major depression

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2002-09; Study Completion 2006-11

PRIMARY OUTCOMES:
Relapse - subject meets criteria for an episode of major depression for 2 weeks or more.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Levitt, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada